CLINICAL TRIAL: NCT03661775
Title: Serum Magnesium Level Between Administered Rate of 2 g/hr Versus 2.5 g/hr in Severe Pre-eclampsia Obese Pregnancy, Multicentered Randomized Study
Brief Title: Serum Magnesium Level Administration in Severe Pre-eclampsia Obese Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: RJMAG001
Record Dates: First submitted 2018-05-14; First posted 2018-09-07 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2018-09

CONDITIONS: Severe Pre-eclampsia; Magnesium Level
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Factorial 2-by-2 open labeled randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- controlled group (Experimental): controlled group : administration of magnesium sulfate is 4 grams for loading dose in 15 minutes, followed by 2 grams for maintenance dose per hour
  Interventions: Drug: Magnesium sulfate administration
- Experimental group (Experimental): group : administration of magnesium sulfate is 4 grams for loading dose in 15 minutes, followed by 2.5 grams for maintenance dose per hour
  Interventions: Drug: Magnesium sulfate administration

INTERVENTIONS:
Drug: Magnesium sulfate administration — controlled group : administration of magnesium sulfate is 4 grams for loading dose in 15 minutes, followed by 2 grams for maintenance dose per hour Experimental group : administration of magnesium sulfate is 4 grams for loading dose in 15 minutes, followed by 2.5 grams for maintenance dose per hour

SUMMARY:
Comparison of the magnesium level in difference continuous rate in women who were diagnosed severe pre-eclampsia obese

DETAILED DESCRIPTION:
Magnesium sulfate is, generally, applied in order to alleviate or to avoid seizures. It can be administered according to many medical approaches. Nevertheless, at Rajavithi Hospital, the recommended administration of magnesium sulfate is 4 grams for loading dose in 15 minutes, followed by 2 grams for maintenance dose per hour (Zudpan regimen). The therapeutic index of magnesium is in the range of 4.8-8.4 mg/dL. After that, the level of magnesium sulfate will be evaluated every 4 or 6 hours.

At Rajavithi Hospital, there are a lot of patients having pre-eclampsia symptom and many patients, who were received magnesium sulfate in the treatment, having the level of magnesium sulfate lower than the therapuetic level and needed to increase the maintenance dose to 2.5 grams/hour. Therefore, this work aims to studying the amount of magnesium sulfate administered to pregnant woman with pre-eclampsia symptom who possess high body mass index (BMI), especially for BMI greater than or equal to 30 kg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy women who have MBI ≥ 31kg/m2
* Pregnancy women who were diagnosed severe pre-eclampsia at gestational age 24 weeks more.
* Pregnancy women who were diagnosed eclampsia at gestational age 24 weeks more.

Exclusion Criteria:

* Pregnancy women who were chronic kidney disease or have serum creatinine more than 1.1 mg/dl
* Pregnancy women who have contraindication to use magnesium sulfate

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
therapeutic level | 4 hours after infusion magnesium sulfate
  Serum magnesium level

SECONDARY OUTCOMES:
Outcome of pregnancy | 24 hours after delivery
  maternal and fetal outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Diaz V, Long Q, Oladapo OT. Alternative magnesium sulphate regimens for women with pre-eclampsia and eclampsia. Cochrane Database Syst Rev. 2023 Oct 10;10(10):CD007388. doi: 10.1002/14651858.CD007388.pub3. PMID 37815037